CLINICAL TRIAL: NCT04540393
Title: A Phase III Open-label Study in Adults to Determine the Safety and Immunogenicity of AZD1222, a Non-replicating ChAdOx1 Vector Vaccine, for the Prevention of COVID-19
Brief Title: AZD1222 Vaccine for the Prevention of COVID-19
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was put on hold in September 2020 due to a safety concern in another trial but never restarted. In the meantime our clinical development program now includes a similar study with a different design, which we prefer to complete now.
Sponsor: AstraZeneca (Industry)
Collaborators: Iqvia Pty Ltd (Industry); Covance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: D8111C00001
Record Dates: First submitted 2020-08-26; First posted 2020-09-07 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: COVID-19
Keywords: COVID-19 Prevention; AZD1222 vaccine for COVID-19 Prevention
MeSH Terms: conditions — COVID-19 | interventions — ChAdOx1 nCoV-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm A (Experimental): Single arm
  Interventions: Biological: AZD1222

INTERVENTIONS:
Biological: AZD1222 — Participants will receive 2 doses of AZD1222; the first dose will be administered on Day 1 and the second dose on Day 29. Unit dose strength(s) > 0.7 × 1011 vp/mL. Dosage level(s) 5 ×1010 vp (nominal). Route of administration Intramuscular injection

SUMMARY:
The purpose of this study is to evaluate safety and immunogenicity of AZD1222 for COVID-19 prevention in the Russian Federation

DETAILED DESCRIPTION:
This is a prospective, multicentre, open-label, non-comparative clinical study, designed to provide data on the use of AZD1222 in the Russian Federation. The protocol is part of the international AstraZeneca program of AZD1222 development with several studies being conducted in the UK, US, Japan, and other countries. This study is intended for registration purposes of AZD1222 in Russia. The study data will complement the data from other pivotal controlled studies conducted in other countries with the Russian participants' data, which is considered the most expedited way to make the severe acute respiratory syndrome-coronavirus-2 (SARS-CoV-2) vaccine available to the Russian Federation for contribution to controlling the current public health crisis.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥ 18 years of age at the time of signing the informed consent.
2. Medically stable such that, according to the judgment of the investigator, hospitalization within the study period is not anticipated and the participant appears likely to be able to remain in follow-up through the end of protocol-specified follow-up.

   * A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months prior to enrolment
3. Able to understand and comply with study requirements/procedures based on the assessment of the investigator.
4. Male and/or female
5. Female participants

   1. Women of childbearing potential must:

      * Have a negative pregnancy test on the day of screening and on Day 1
      * Use one highly effective form of birth control for at least 28 days prior to Day 1 and agree to continue using one highly effective form of birth control through 60 days following administration of the second dose of study intervention. A highly effective method of contraception is defined as one that can achieve a failure rate of less than 1% per year when used consistently and correctly. Periodic abstinence, the rhythm method, and withdrawal are NOT acceptable methods of contraception.
   2. Women are considered of childbearing potential unless they meet either of the following criteria:

      * Surgically sterilised (including bilateral tubal ligation, bilateral ophorectomy, or hysterectomy), or
      * Postmenopausal
      * For women aged < 50 years, postmenopausal is defined as having both:

        * A history of ≥ 12 months amenorrhea prior to first dosing, without an alternative cause, following cessation of exogenous sex-hormonal treatment, and
        * A follicle-stimulating hormone level in the post-menopausal range Until follicle-stimulating hormone is documented to be within menopausal range, the participant is to be considered of childbearing potential
      * For women aged ≥ 50 years, postmenopausal is defined as having a history of ≥ 12 months amenorrhea prior to first dosing, without an alternative cause, following cessation of exogenous sex-hormonal treatment
6. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in the protocol

Exclusion Criteria:

1. History of allergic disease or reactions likely to be exacerbated by any component of AZD1222.
2. Active infection with SARS-CoV-2 as confirmed by RT-PCR.
3. Known past laboratory-confirmed SARS-CoV-2 infection. Note: Participant's baseline serostatus determined as part of the study will not be used as a basis for exclusion from the study.
4. Significant infection or other acute illness, including fever > 37.8°C on the day prior to or day of first dosing.
5. Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent severe infections and use of immunosuppressant medication within the past 6 months (≥ 20 mg/kg/day of prednisone or its equivalent, given daily or on alternate days for ≥ 15 days within 30 days prior to administration of study intervention), except topical/inhaled steroids or short-term oral steroids (course lasting

   ≤ 14 days).
   1. Note: HIV-positive participants with CD4 counts > 500 for ≥ 12 months and on a stable HIV antiretroviral regimen may be enrolled
   2. Note: Topical tacrolimus is allowed if not used within 14 days prior to the day of erolment.
6. History of primary malignancy except for:

   1. Malignancy with low potential risk for recurrence after curative treatment (for example, history of childhood leukaemia) or metastasis (for example, indolent prostate cancer) in the opinion of the site investigator.
   2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   3. Adequately treated uterine cervical carcinoma in situ without evidence of disease
   4. Localised prostate cancer
7. Clinically significant bleeding disorder (eg, factor deficiency, coagulopathy, or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture.
8. Severe and/or uncontrolled cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, and neurological illness, as judged by the investigator (mild/moderate well-controlled comorbidities are allowed).
9. History of Guillain-Barré syndrome, or other neuroimmunological disease.
10. Any other significant disease, disorder, or finding that may significantly increase the risk to the participant, affect the ability of the participant to participate in the study, or impair interpretation of the study data.
11. Receipt of, or planned receipt of investigational products indicated for the treatment or prevention of SARS-CoV-2 or COVID-19. Note: For participants in the study who become hospitalised with COVID-19, receipt of licensed treatment options and/or participation in investigational treatment studies is permitted.
12. Receipt of any vaccine (licensed or investigational) other than licensed influenza vaccines within 30 days prior to and after administration of study intervention.
13. Receipt of any influenza vaccine (licensed or investigational) within 7 days prior to and after administration of study intervention.
14. Receipt of immunoglobulins and/or any blood products within 3 months prior to administration of study intervention or expected receipt during the period of study follow-up.
15. Involvement in the planning and/or conduct of the study (applies to both Sponsor staff and/or staff at the study site).
16. For women only - currently pregnant (confirmed with positive pregnancy test) or breastfeeding
17. Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.
18. Previous enrolment in the present study. 5.3 Lifestyle Considerations 1) Participants must follow the contraception requirements 2) Restrictions relating to concomitant medications

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2020-12-04 (Estimated); Study Completion 2022-05-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of SAEs following the first vaccination and throughout the study duration (Day 180) [Safety and Tolerability]. | 180 days
  Occurrence of SAEs following the first vaccination and throughout the study duration (Day 180).

SECONDARY OUTCOMES:
Incidence of Solicited AEs for 7 following each vaccination [Safety and Tolerability]. | 180 days
  Local and systemic solicited AEs for 7 days following each vaccination. Unsolicited AEs for 28 days following each vaccination.
  Occurrence of AESIs following the first vaccination and throughout the study duration (Day 180).
SARS-CoV-2 antigen-specific antibody levels | 180 days
  immunogenicity / serologic responses to AZD1222
The rate of participants seroconverting from negative to positive SARS-CoV-2 S antigen | 180 days
  immunogenicity / serologic responses to AZD1222
The rate of participants seroconverting from negative to positive SARS-CoV-2 N | 180 days
  immunogenicity / serologic responses to AZD1222
Quantity of SARS-CoV-2 neutralizing antibodies | 180 days
  immunogenicity / serologic responses to AZD1222
Count of peripheral blood mononuclear cells (PBMCs) | 180 days
  immunogenicity / serologic responses to AZD1222
Quantity of seasonal coronavirus antigens | 180 days
  immunogenicity / serologic responses to AZD1222
Quantity of antibodies to the ChAdOx1vector and the persistence of these antibodies over time | 180 days
  immunogenicity / serologic responses to AZD1222

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home